CLINICAL TRIAL: NCT03653572
Title: Clinical Evaluation of the Next Generation Venue Ultrasound System, Components, and Accessories - Canada
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 110.04-2016-GES-0007
Record Dates: First submitted 2018-01-22; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Ultrasound Use in Emergency/Medical Care
Keywords: Ultrasound; Emergency care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Eligible Subjects (Other): All subjects will be enrolled into a single arm and will undergo an ultrasound exam, per the protocol.
  Interventions: Device: Ultrasound exam

INTERVENTIONS:
Device: Ultrasound exam — Eligible subjects will be positioned for their ultrasound exam, which will take a similar amount of time and be performed in a similar manner as standard of care ultrasound exams at the site. The type and duration of ultrasound exam will be based on the subject's clinical condition.

SUMMARY:
The purpose of the study is to collect images data sets from clinical cases and periodic user feedback on the Next Generation Venue ultrasound system under clinical conditions. This is a medical device study designed as a clinical, open label, unblinded, non-randomized, prospective, feasibility research study.

DETAILED DESCRIPTION:
Adult patients (aged >18 years) will be enrolled as they present for emergency or immediate medical care, in facilities such as the intensive care unit (ICU), cardiac care unit (CCU), and/or other departments. Subjects may or may not have a clinical indication for ultrasound scanning as part of their regular medical care and will be required to meet the inclusion criteria and none of the exclusion criteria. Eligible subjects will undergo an ultrasound exam using the investigational ultrasound device. The exam type will be based on the subject's clinical condition. Users performing the scans will periodically be asked to provide feedback on User Survey forms prepared by the Sponsor. Image data sets from investigational exam will be stored electronically and de-identified data will be disclosed to the Sponsor.Results are for use in development and optimization of a next generation ultrasound system being developed by study Sponsor, GE Healthcare (GEHC) prior to future commercial release.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (aged 18 years of age or older) at the time of consent;
2. Eligible to undergo ultrasound scanning per the site standard of care (with or without a clinical indication for scanning); AND
3. Able and willing to provide written informed consent for participation.

Exclusion Criteria:

1. Are pregnant subjects;
2. Require procedures that cannot be readily completed using available investigational devices; OR
3. Require or are anticipated to require medical care where study participation could reasonably be expected to adversely impact patient care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Obtain Image sets using Ultrasound Venue System | Two months
  Number of representative image sets for subjects enrolled in study
Periodic user feedback | Two months
  Periodic user feedback data from device users.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Girard, MD, Principal Investigator — Hopital Notre-Dame
Locations (1):
- Hopital Notre-Dame, Montreal, Quebec, Canada